CLINICAL TRIAL: NCT04690153
Title: Novel Approach of Hayman Uterine Compression Sutures for Management of Severe Atonic Postpartum Hemorrhage: Three Vertical Sutures
Status: Completed | Type: Observational
Sponsor: Pınar Yalcin bahat (Other)
Collaborators: Ismail Ozdemir (Unknown)
Responsible Party: Sponsor-Investigator, Pınar Yalcin bahat, Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: hayman
Record Dates: First submitted 2020-12-19; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Uterine Atony
MeSH Terms: conditions — Uterine Inertia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with three vertical Hayman Sutures — Patients who are referred to our clinic due to postpartum hemorrhage between the ages of 18-45 and who need to undergo a surgical procedure (not responding to medical treatment) due to abnormal uterine bleeding in our clinic will be included. Patients with a previously known diagnosis of bleeding and coagulation disorders will not be included in the study. Considering that we are one of the primary referral centers in Istanbul in terms of deliveries and post-partum bleeding in our hospital, it is aimed to terminate the study with approximately 50 participants.

SUMMARY:
Maternal deaths due to uterine atony bleeding are the leading causes of maternal death in our country and all over the world. In this respect, our clinic is among the clinics with the highest number of experience in our country and aims to reduce maternal deaths and mothers who will need intensive care due to bleeding with a hemorrhage stopping technique that will have a serious contribution to both our country and the world literature.

Our primary goal, thanks to the bleeding-stopping technique, to reduce their deaths. Our secondary aim is, thanks to the bleeding-stopping technique we offer, To prevent and reduce the complications seen in mothers during the operative period.

DETAILED DESCRIPTION:
Our research was carried out to our obstetrics clinic between 01 Agustus 2015 - 01 December 2020.

Patients transplanted due to postpartum bleeding and patients requiring surgery due to abnormal postpartum bleeding in our clinic will be included. Patients with a previously known bleeding disorder will not be included in the study. In our study, the parameters of the patients who had bleeding due to postpartum uterine atony and who needed uterine surgery previously underwent triple Hayman compression suture to stop bleeding will be included in the study. Patients with a triple Hayman suture covering the upper 2/3 of the uterus to stop uterine bleeding will be evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum bleeding after birth
* Patients referred to our clinic from an external center due to postpartum bleeding
* Patients who have given birth due to pregnancy older than 24 weeks and have atony bleeding

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients with abnormal uterine bleeding other than birth Patients with known metabolic diseases Patients with known bleeding and coagulation disorders
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Reduce maternal deaths due to bleeding | 5 years
  Maternal death due to uterine atony is common all over the world, especially in developing countries. Thanks to the technique we apply, it is aimed to reduce bleeding and decrease maternal deaths.

SECONDARY OUTCOMES:
to prevent and reduce complications seen in mothers in the post-operative period due to bleeding, | 5 years
  Some complications may occur due to excessive bleeding after uterine atony. These complications can be permanent or fatal. (for example, acute renal failure, disseminated intravascular coagulation disorder, etc., it is aimed to reduce these with the applied technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No